CLINICAL TRIAL: NCT01568788
Title: Post-marketing Clinical Observation of Hualan's Inactivated Influenza Vaccine: A Single Center, Parallelled, Controlled, Randomised Clinical Trial
Brief Title: Post-marketing Clinical Observation of an Inactivated Influenza Split Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hualanbio-influenza-IV-002; Hualanbio-003 (Other Grant/Funding Number: Hualan Biological Engineering INC.)
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-04

CONDITIONS: Human Influenza
Keywords: Respiratory Tract Infections; Orthomyxoviridae Infections
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections; Orthomyxoviridae Infections | interventions — vaxigrip; fluarix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inactivated Influenza Vaccine (Experimental): 15μg HA/strain/0.5ml/syringe, Hualan Biologicals
  Interventions: Biological: Inactivated Influenza Vaccine
- Inactivated Influenza Vaccine of Pasteur (Active Comparator): 15ug HA/strain/0.5ml/syringe, Sanofi Pasteur
  Interventions: Biological: Inactivated Influenza Vaccine of Pasteur
- Inactivated Influenza Vaccine of GSK (Active Comparator): 15ug HA/strain/0.5ml/syringe, GSK
  Interventions: Biological: Inactivated Influenza Vaccine of GSK

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine — 200 subjects were randomly assigned (60 children, 100 adults and 40 elders) to receive Inactivated Influenza Vaccine (Split virion) of Hualan Biologicals, 15ug HA/strain/0.5ml/syringe, one dose regime
  Other Names: Hualan Biologicals
  Arms: Inactivated Influenza Vaccine
Biological: Inactivated Influenza Vaccine of Pasteur — 200 subjects (60 children, 100 adults and 40 elders) were randomly assigned to receive the Inactivated Influenza Vaccine of Sanofi Pasteur, 15ug HA/strain/0.5 ml/syringe, one dose regime,
  Other Names: VAXIGRIP
  Arms: Inactivated Influenza Vaccine of Pasteur
Biological: Inactivated Influenza Vaccine of GSK — 200 subjects (60 children, 100 adults and 40 elders) were randomly assigned to receive Inactivated Influenza Vaccine (Split virion) of GSK, 15ug HA/strain/0.5ml/syringe, one dose regime
  Other Names: Fluarix
  Arms: Inactivated Influenza Vaccine of GSK

SUMMARY:
Phase III clinical trial was carried out in Jintan city, Jiangsu Province, China in May, 2006. Trial results showed that the vaccine had proved safety and immunogenicity. Influenza vaccine of Hualanbio has obtained production permission and marketing authorization in May, 2008.

In order to further investigate the safety and immunogenicity of the vaccine in the market, The clinical observation was planned to be conducted in Mianyang city (Yanting County), Sichuan Province, China.

DETAILED DESCRIPTION:
Dosage and administration route in this clinical trial:

Subjects age 3 years or older was vaccinated following a single 0.5ml dose immunization regime.

The preferred site of injection was the at the skin near outboard deltoid muscle of the upper arm.

The administration route is after the sanitization with 75% alcohol, intramuscularly inject the test vaccine or the control vaccines when the skin was slightly dried for those subjects complied with the inclusion requirements.

Safety indicators:

* Post-vaccination local and systemic adverse reaction levels, together with the soliciting adverse reaction within 30 minutes ;
* Post-vaccination local and systemic adverse reaction levels, together with the soliciting adverse reactions through 6 hours to the 29th day ;
* Summarize the adverse events/severe adverse events and the incidence levels from the inclusion of the subjects to the completion of the clinical trial.

Immunogenicity indicators:

Evaluate the Post-vaccination immunogenicity of the test and the control influenza vaccines in persons age 3 years and older by its HI antibody level on Day 28.

Take 1:10 serum dilution as the minimum dilutability. The seroconversion in this trial was defined as the post-vaccination HI antibody titer ≥ 1:40 when the HI antibody < 1:10 before the vaccination or the post-vaccination HI antibody titer quadruply increased when HI antibody ≥ 1:10 before the vaccination.

The Immunogenicity criteria set for this clinical trial is the seroconversion shall be > 40% after 14 days of the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female age 3 and older, volunteers or their guardians are able to understand and sign the informed consent;
* Healthy male or female by inquiring illness history, physical examination and clinical judgment and who complies with vaccination of this product;
* Be able to comply with the requirement of clinical trial protocol;
* Have no history of vaccination within the past 6 months and vaccination with other product within the latest 1 week;
* Axillary temperature <37.1℃.

Exclusion Criteria:

* Subject that was allergic to eggs and any component of the vaccine, or has history of other allergy;
* Fever, acute disease or acute onset of chronic disease and influenza;
* Guillain-Barre Syndrome

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse reactions as a measure of safety study | 28 days after the vaccination
  Local reactions, systemic reactions, severity degree and AEFI correlation

SECONDARY OUTCOMES:
Observation of the immunological effect | 28 days after the immunization
  HI antibody seroconversion ratios

CONTACTS AND LOCATIONS:
Overall Officials: Pei-ru Zhang, Principal Investigator — Immune Planning Institute of Mianyang Center for Disease Prevention and Control
Locations (1):
- Yanting County, Mianyang, Sichuan, China

REFERENCES:
- [Result] Zhang PR, Zhu XP, Zhou LJ, Liu YQ, Fan Y, Chen G, Chen Z, Liu Y, Sun HY, Wu JL. [Safety and immunological effect of domestic split influenza virus vaccine]. Zhonghua Yu Fang Yi Xue Za Zhi. 2009 Jul;43(7):615-8. Chinese. PMID 19954075